CLINICAL TRIAL: NCT01019538
Title: COPD and Air Travel: Oxygen Equipment and Pre-flight Titration of Supplemental Oxygen
Brief Title: Pre-flight Titration of Supplemental Oxygen
Status: Completed | Type: Observational
Sponsor: Ullevaal University Hospital (Other)
Responsible Party: Ole Henning Skjønsberg, Prof., dr.med, Oslo University Hospital, Ullevaal, Department of Pulmonary Medicine
Organization: Oslo University Hospital (Other)
Other Study IDs: 897
Record Dates: First submitted 2009-11-23; First posted 2009-11-25 (Estimated); Last update posted 2011-07-06 (Estimated); Status verified 2009-11

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Oxygen; Hypoxemia; Air travel
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Hypoxia | interventions — Oxygen

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Arterial blood gases
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: Pre-flight test with supplemental oxygen — The Hypoxia-altitude simulation test, which is established in clinical practice, is compared to the gold standard of hypobaric chamber while giving supplemental gaseous oxygen without and with oxygen conserving device, and with oxygen concentrator.
  Other Names: Oxygen

SUMMARY:
The purpose of this study is to evaluate if supplemental oxygen during air travel can be reliably titrated using a Hypoxia-altitude simulation test (HAST). Also, the effect of oxygen supplementation given with the various oxygen equipment allowed for air travel is studied.

DETAILED DESCRIPTION:
International guidelines recommend supplemental oxygen if PaO2 < 6.7 kPa (50 mmHg) during air travel. Hypobaric chamber exposure is the ideal test but is not widely available. In clinical practice, the HAST has been recommended as the preferable test for pre-flight evaluation, and is used with increasing frequency. The oxygen dose during air travel has been recommended titrated during HAST. In the study, supplemental oxygen titration during hypobaric chamber exposure is compared to oxygen titration during HAST, to evaluate if HAST can be used with confidence to titrate the amount of supplemental oxygen needed during air travel.

ELIGIBILITY:
Inclusion Criteria:

* COPD patients who have performed a Hypoxia-altitude simulation test with a PaO2 < 6.7 kPa

Exclusion Criteria:

* exacerbation or pneumothorax within the previous six weeks
* LTOT
* anemia
* pulmonary disease other than COPD
* cerebrovascular or symptomatic cardiovascular disease
* claustrophobia
* inability to equalize pressure in the middle ear

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: COPD patients
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2008-12; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
PaO2 obtained from oxygen titration during HAST vs hypobaric chamber | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Ole H Skjønsberg, Prof.dr.med, Study Director — Oslo University Hospital; Aina Akerø, M.D., Principal Investigator — Oslo University Hospital
Locations (1):
- Oslo University Hospital Ullevaal, Department of Pulmonary Medicine, Oslo, Oslo County, Norway

REFERENCES:
- [Background] Gong H Jr, Tashkin DP, Lee EY, Simmons MS. Hypoxia-altitude simulation test. Evaluation of patients with chronic airway obstruction. Am Rev Respir Dis. 1984 Dec;130(6):980-6. doi: 10.1164/arrd.1984.130.6.980. PMID 6508019
- [Background] Akero A, Christensen CC, Edvardsen A, Skjonsberg OH. Hypoxaemia in chronic obstructive pulmonary disease patients during a commercial flight. Eur Respir J. 2005 Apr;25(4):725-30. doi: 10.1183/09031936.05.00093104. PMID 15802350
- [Background] Akero A, Christensen CC, Edvardsen A, Ryg M, Skjonsberg OH. Pulse oximetry in the preflight evaluation of patients with chronic obstructive pulmonary disease. Aviat Space Environ Med. 2008 May;79(5):518-24. doi: 10.3357/asem.2120.2008. PMID 18500050
- [Background] Dine CJ, Kreider ME. Hypoxia altitude simulation test. Chest. 2008 Apr;133(4):1002-5. doi: 10.1378/chest.07-1354. PMID 18398121
- [Derived] Akero A, Edvardsen A, Christensen CC, Owe JO, Ryg M, Skjonsberg OH. COPD and air travel: oxygen equipment and preflight titration of supplemental oxygen. Chest. 2011 Jul;140(1):84-90. doi: 10.1378/chest.10-0965. Epub 2010 Nov 11. PMID 21071527